CLINICAL TRIAL: NCT07202221
Title: Evaluation of Spoken Animation as a Tool for Imparting Information About Epidural Labour Analgesia
Brief Title: Spoken Animation for Labour Epidural
Acronym: SALE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chelsea and Westminster NHS Foundation Trust (Other)
Collaborators: Imperial College London (Other); University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 351150-SALE; 351150 (Other: NIHR)
Record Dates: First submitted 2025-06-19; First posted 2025-10-01 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Labour Pain
Keywords: labour; consent; information; animation; obstetric; epidural
MeSH Terms: conditions — Labor Pain

STUDY DESIGN:
Intervention Model Description: Participants randomly assigned to one of two groups for comparative analysis.
Masking Description: Masking is not possible as the intervention involves the addition of an animated film, which is not seen by the control group. The patient and the investigator are therefore inherently aware of the randomly assigned study group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): Participant receives written information about epidural alone
  Interventions: Other: Participant receives current gold standard written information alone
- Intervention group (Experimental): Participant receives animated introductory film in addition to written information about epidural
  Interventions: Other: Participant views Epidural animation before reading gold standard written information

INTERVENTIONS:
Other: Participant views Epidural animation before reading gold standard written information — Addition of introductory animation to written OAA epidural information card about labour epidural
  Arms: Intervention group
Other: Participant receives current gold standard written information alone — Gold standard OAA (Obstetric Anaesthetists' Association) epidural information card
  Arms: Control group

SUMMARY:
The purpose of this study is to evaluate a new animated information film as a tool for introducing the concept of epidural as a method of labour pain relief to expectant women.

The main question that the study is designed to answer is:

Compared to written information alone, does the addition on a short animated introductory film reduce decisional conflict for expectant women regarding the use of epidural pain relief.

Secondary outcomes tested will be change in anxiety and satisfaction scores after receiving the information.

Study participants will include women expecting their first baby, presenting to hospital for induction of labour. They will be asked to fill out a questionnaire regarding thoughts and feelings around epidural, before and after receiving information about the procedure. Participants will be randomised to receive either traditional written information alone or with the addition of the animated film.

A smaller number of participants will also be asked to participate in a short interview about the animated film.

DETAILED DESCRIPTION:
This study is a prospective, randomised controlled trial with a pre-post design, as well as a qualitative analysis of user acceptability.

The planned sample size is 60 in control group, 60 in intervention group (120 in total). The study will only involve primiparous women presenting to the antenatal ward for induction of labour.

Participation in the study will take place on the antenatal unit, before transfer to labour ward. Participants will be asked to complete a pre-intervention survey regarding decisional conflict score for labour analgesia choices and including Likert scales for anxiety and understanding related to epidural.

They will then be given information about epidural for labour analgesia - the control group will receive written information alone; the intervention group will watch a short animation introducing the concept of epidural, followed by the same written information.

This will be followed by a post-intervention survey. A smaller group will be selected (dependent on availability of interviewer) for a short interview to allow qualitative analysis of the acceptability and effectiveness of the animation.

ELIGIBILITY:
Inclusion Criteria:

• Primiparous birthing people presenting for induction of labour.

Exclusion Criteria:

* Patient refusal
* Unable to speak English or any of the seven language translations provided
* Epidural contraindicated
* Previous Epidural for any reason
* Any significant health concerns

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-10-15 (Estimated); Primary Completion 2026-10-15 (Estimated); Study Completion 2026-10-15 (Estimated)

PRIMARY OUTCOMES:
Change in Decisional Conflict Score | Day 1
  Change in total Decisional Conflict Score (DCS) regarding labour epidural, before and after exposure to information material.
  The DCS is measured by response to various statements on a five point Likert scale: Maximum value = strongly agree, minimum value = strongly disagree. Strongly agree responses represent a better outcome.

SECONDARY OUTCOMES:
Change in the following DCS subscore categories. | Day 1
  Change in the following DCS subscore categories: uncertainty, informed, values clarity, support, effective decision.
  The DCS is measured by response to various statements on a five point Likert scale: Maximum value = strongly agree, minimum value = strongly disagree. Strongly agree responses represent a better outcome.
Self-reported Likert scale outcomes | Day 1
  Self-reported Likert scale outcomes for understanding of the epidural procedure, associated anxiety and overall satisfaction with information received.
  Scale: Five point Likert scale; Maximum value = strongly agree, minimum value = strongly disagree. Strongly agree responses represent a better outcome, with one exception where the minimum value means a better outcome (response to statement: "I feel anxious about the idea of having an epidural")

OTHER OUTCOMES:
Qualitative analysis of post intervention structured interviews. | Day 1
  Focussed qualitative interviews involving a smaller patient group - to assess acceptability and specific feedback for the animated film itself.

CONTACTS AND LOCATIONS:
Overall Officials: Charles Prior, FRCA, Principal Investigator — Chelsea & Westminster NHS Trust
Locations (1):
- West Middlesex Hospital, Chelsea & Westminster NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-03-12): https://cdn.clinicaltrials.gov/large-docs/21/NCT07202221/Prot_SAP_000.pdf
  • Informed Consent Form (2025-03-12): https://cdn.clinicaltrials.gov/large-docs/21/NCT07202221/ICF_001.pdf